CLINICAL TRIAL: NCT01826123
Title: Point-of-Care Testing - A Prospective, Randomized, Controlled Multicenter Study of Efficacy in Coagulopathic Cardiac Surgery Patients
Brief Title: Point-of-Care Testing in Coagulopathic Patients Undergoing Cardiac Surgery - a Multicenter Study
Acronym: MultiPOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Christian F. Weber, MD, Dr. med. Dr. med. habil. Christian Friedrich Weber, Goethe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 343/12
Record Dates: First submitted 2013-03-19; First posted 2013-04-08 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Coagulopathy During Cardiac Surgery
Keywords: Coagulopathy; Hemorrhage; Cardiac surgery; Point-of-Care testing; POC; ROTEM; multiplate; Multiple electrode aggregometry (MEA)
MeSH Terms: conditions — Hemostatic Disorders; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional laboratory testing (Active Comparator): After being randomized to the group "conventional coagulating testing", hemostatic therapy will be based exclusively on conventional standard coagulation analyses like International normalized ratio (INR), activated prothrombin time (aPTT), fibrinogen and platelet concentration or Activated clotting time (ACT. Analyses will be performed at i) fixed time points (preoperative and at admission to ICU) and ii) variable timepoints depending on the decision of the attending physician. Hemostatic therapy will be based on a specific hemostatic therapy algorithm. Intraoperatively, analyses of ACT (activated clotting time) and INR will be performed following institutional standards using specific POC tests.
  Interventions: Device: Conventional laboratory testing (Central laboratory)
- POC testing (ROTEM and Multiplate) (Active Comparator): After being randomized to the group "POC testing", hemostatic therapy will be based exclusively on POC measures obtained by i) viscoelastic tests (ROTEM(R), TEM international, Munich, Germany) and aggregometric tests (multiplate, ROCHE AG, Grenzach, Germany). Analyses will be performed at variable timepoints depending on the decision of the attending physician. Hemostatic therapy will be based on a specific hemostatic therapy algorithm. Intraoperatively, analyses of ACT (activated clotting time) and INR will be performed following institutional standards using specific POC tests.
  Interventions: Device: POC testing

INTERVENTIONS:
Device: Conventional laboratory testing (Central laboratory) — aPTT, INR, fibrinogen concentration, platelet count
  Arms: Conventional laboratory testing
Device: POC testing — ROTEM: Clotting time (CT) in the EXTEM- and INTEM-test, Maximal clot firmness in the FIBTEM-test, Clot Lysis Index (CLI) multiplate: Area under the aggregation curve following stimulation with arachidonic acid (ASA) and Adenosine diphosphate (ADP)
  Other Names: viscoleastic measures using the ROTEM(R) device and; aggregometric measures using the Multiplate(R) device
  Arms: POC testing (ROTEM and Multiplate)

SUMMARY:
Recently, the investigators study group showed in a mono center study that Point of Care (POC) based hemotherapy may reduce transfusion rates of allogenic blood products in perioperative care of coagulopathic cardiac surgery patients. The investigators aim to verify the obtained results by conducting this multicenter study.

ELIGIBILITY:
Inclusion Criteria:

Step 1:

* Patients scheduled for elective, complex cardiothoracic surgery (combined coronary artery bypass graft and valve surgery, double or triple valve procedures, aortic surgery or redo surgery) with cardiopulmonary bypass (CPB)

Step 2:

* diffuse bleeding after heparin reversal following extracorporeal circulation or
* intra- or postoperative blood loss exceeding 250 ml/h or 50 ml/10 min

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-07; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
packed red blood cell concentrate (PRBC) transfusion rate | During the period between inclusion into the study and 24 h after postoperative admission to ICU
  Number of transfused units of PRBC during the period between inclusion into the study and 24 hours (h) after admission to ICU.

SECONDARY OUTCOMES:
Transfusion rate of Fresh Frozen Plasma | During the period between inclusion into the study and 24 h after postoperative admission to ICU
  Number of transfused units of Fresh Frozen Plasma (FFP)
Postoperative Blood loss | for up to 24 h after postoperative admission to ICU
  Blood loss 6h, 12h and 24h after postoperative admission to ICU
Duration of mechanical ventilation | after postoperative admission to ICU, an expected average of 30 hours
  Duration of postoperative mechanical ventilation
Horovitz - indices | for up to 24 h after postoperative admission to ICU
  PaO2/FiO2 - indices at admission to ICU, as well as 2h, 4h, 12h and 24 h after admission to ICU
Incidence of acute renal failure | during treatment at the intensive care unit, for an average of 3 weeks
  Incidence of acute renal failure
Duration of hospitalisation | From admission to ICU and up to discharge from the hospital, an expected average of 10 days
  duration of ICU treatment duration of IMC (Intermediate Care) treatment duration of hospitalisation
rethoracotomies | During the period between inclusion into the study and 24 h after postoperative admission to ICU
  number of patients with rethoracotomies. Cause for rethoracotomies (surgical or coagulopathic bleeding, pericardium tamponade)
Thromboembolic or allergic adverse events | for up to 24 h after postoperative admission to ICU
  Number of patients with thromboembolic or allergic adverse events.
Ventilator - associated pneumonia | after postoperative admission to ICU up to discharge from ICU, an expected average of 5 days
  Number of patients with ventilator - associated pneumonia
Postoperative Sepsis | after postoperative admission to ICU up to discharge from ICU, an expected average of 5 days
  Number of patients with postoperative Sepsis
Transfusion rate of platelet concentrates | During the period between inclusion into the study and 24 h after postoperative admission to ICU
  Number of transfused platelet concentrates
Age of each platelet concentrate | During the period between inclusion into the study and 24 h after postoperative admission to ICU
  age (days) of each platelet concentrates
Amount of infused PCC | During the period between inclusion into the study and 24 h after postoperative admission to ICU
  Amount of infused prothrombin complex concentrates (PCC)
Amount of infused rVIIa | During the period between inclusion into the study and 24 h after postoperative admission to ICU
  Amount of infused activated coagulation factor VII (rVIIa)
Amount of infused fibrinogen concentrate | During the period between inclusion into the study and 24 h after postoperative admission to ICU
  Amount of infused fibrinogen concentrate

OTHER OUTCOMES:
Preoperative antiaggregatory medication | at the day before surgery
  number of patients with preoperative intake of any antiaggregatory medication. kind of antiaggregatory medication.
infused crystalloid and colloid volume | intraoperatively and for up to 24 h after admission to ICU
  Amount of infused crystalloid and colloid volume. kind of crystalloid and colloid volume.
Age | at the day before surgery
  age of the patient
euroSCORE | at the day before surgery
  perioperative risk assessment
Weight | at the day before surgery
  Weight of the patient
Height | at the day before surgery
  height of the patient
ASA score | at the day before surgery
  Preoperatively assessed anesthesia risk score
clamping time | intraoperatively
  Duration of intraoperative clamping of the aorta
CPB time | intraoperatively
  Duration of extracorporeal circulation intraoperatively
Priming volume | intraoperatively
  Volume of the priming volume of the extracorporeal circulation
INR | preoperatively and up to 24 h after admission to ICU
  International Normalized Ratio
aPTT | preoperatively and up to 24 h after admission to ICU
  activated partial prothrombin time [sec]
Platelet count | preoperatively and up to 24 h after admission to ICU
  platelet count
CT | Intraoperatively and up to 24 h after admission to ICU
  Clotting time in the EXTEM and INTEM test of the Rotem device
MCF | intraoperatively and up to 24h after admission to ICU
  Maximal clot firmness in the EXTEM- and INTEM test of the ROTEM device
AUC | intraoperatively and up to 24h after admission to ICU
  Area under the aggregation curve in the Multiplate device following stimulation with arachidonic acid or adenosine disphosphate.

CONTACTS AND LOCATIONS:
Overall Officials: Christian F Weber, MD, Study Director — Goethe University; Kai Zacharowski, PhD, MD, Principal Investigator — Goethe University; Alexander Schellhaaß, MD, Study Chair — Heidelberg University; Stefan Hofer, PhD, MD, Study Chair — Heidelberg University; Roland Freynschlag, MD, Study Chair — University of Linz; Hans Gombotz, PhD, MD, Study Chair — University of Linz; Jan Roesner, MD, Study Chair — University of Rostock
Locations (4):
- University of Linz, Linz, Upper Austria, Austria
- Germany (3):
  - University of Heidelberg, Heidelberg, Baden-Wurttemberg
  - Goethe - University, Frankfurt am Main, Hesse
  - University of Rostock, Rostock, Mecklenburg-Vorpommern

REFERENCES:
- [Background] Weber CF, Gorlinger K, Meininger D, Herrmann E, Bingold T, Moritz A, Cohn LH, Zacharowski K. Point-of-care testing: a prospective, randomized clinical trial of efficacy in coagulopathic cardiac surgery patients. Anesthesiology. 2012 Sep;117(3):531-47. doi: 10.1097/ALN.0b013e318264c644. PMID 22914710
- [Background] Weber CF, Zacharowski K. Perioperative point of care coagulation testing. Dtsch Arztebl Int. 2012 May;109(20):369-75. doi: 10.3238/arztebl.2012.0369. Epub 2012 May 18. PMID 22685493